CLINICAL TRIAL: NCT04459910
Title: Medial and Lateral Combined Ligament Arthroscopic Repair for Multidirectional Ankle Instability: Case Series
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Nacime Salomão Barbachan Mansur, MD, PhD, Federal University of São Paulo
Other Study IDs: Multi_EPM
Record Dates: First submitted 2020-07-02; First posted 2020-07-07 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Ankle Injuries; Ligament Injury; Joint Instability; Deltoid Ligament; Sprain (Strain) (Ankle); Talofibular Ligament Tear
MeSH Terms: conditions — Ankle Injuries; Joint Instability; Sprains and Strains

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multidirectional: Arthroscopic lateral ligament repair combined with deltoid arthroscopic ligament repair.
  Interventions: Procedure: Arthroscopic Brostrom combined with Arthroscopic Deltoid Repair

INTERVENTIONS:
Procedure: Arthroscopic Brostrom combined with Arthroscopic Deltoid Repair — After anesthesia and surgical site preparation, traditional arthroscopic portals were performed. A 4.5mm set was used to clean the joint and assess possible associated injuries. Anterolateral and anteromedial impacts were resected when needed. Lateral and medial instability were confirmed arthroscopically, and ligament repairs prepared, starting by the lateral compartment. A traditional Arthroscopic Brostrom was performed, using one anchor and suture passers. Sutures are passed but not tightened. Medial anchor insertion is executed at the medial malleolus, in the quadrant described by Vega et al. Sutures were passed respecting the safe zone illustrated by Acevedo at al. The ankle was positioned in neutral (no posterior drawer) and the lateral sutures tightened with arthroscopic knots. Finally, the medial repair is finalized by tightening the deltoid sutures with the ankle at the same position. Portals were closed and a dressing applied.

SUMMARY:
Abstract Introduction: The high prevalence of sprains in the population has provided a substantial number of patients with lateral instability of the ankle. The continuity of this condition can lead to the progressive loosening of the medial containment structures, generating a multidirectional rotational instability. The deltoid approach through the imbrication of its components has been proposed as a solution for these patients. The arthroscopic technique has been described as an alternative.

Methods: This is a retrospective study with patients diagnosed with multidirectional instability and submitted to an ankle arthroscopy with medial repair (arthroscopic tensioning) and lateral (arthroscopic Brostrom) between January 2018 and January 2020. All patients will fill an epidemiological questionnaire and will be evaluated for pain and function according to the Visual Analogue Scale (VAS) and the American Orthopaedic Foot and Ankle Society Score (AOFAS) at 12 months (6-24 months) average of follow-up.

Discussion: The combined medial and lateral arthroscopic repair may be an effective and safe alternative in the treatment of multidirectional instability. The inclusion of the deltoid complex and the low invasiveness of this technique can improve the clinical outcomes of these patients. Additional studies, with a prospective and comparative methodology are required to sustain this proposal.

Design: Level IV. Retrospective case series.

Keywords: ankle injuries; lateral ligament; collateral ligaments; joint instability

ELIGIBILITY:
Inclusion Criteria:

* complaints about ankle loosening for the last six months
* clinical findings of lateral and medial instability

Exclusion Criteria:

* existence of previous surgery
* autoimmune diseases
* neuropathy
* inflammatory disease
* isolated medial instability
* flatfoot
* previous ankle infiltration
* radiographic findings of ankle arthritis
* cavovarus deformity
* coagulopathies
* body mass index over 35
* associated injuries, such as osteochondral lesions
* syndesmosis instability
* tendon ruptures
* fractures

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Tertiary teaching hospital patients, athletes and non-athletes.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
American Orthopedic Foot and Ankle Society - Hindfoot Score (AOFAS) | 6th post-operataive month
  Functional Score (0 to 100 | 100 best score possible | 0 worst score possible)

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | 6th post-operataive month
  Pain Score (0 to 10 | 10 worst score possible | 0 best score possible)
Complications | 6th post-operataive month
  Surgical complications

CONTACTS AND LOCATIONS:
Overall Officials: Nacime Salomão Barbachan Mansur, MD, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
According to the ICMJE data sharing police, core records will be shared at an online depository and available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the article is published.
Access Criteria: A formal requisition will be needed, directly addressed to the main researcher. A good scientific reason must be included.